CLINICAL TRIAL: NCT05848050
Title: Evaluation of the Humoral and Tumoral Molecular Alteration Profile of Brain Metastases
Acronym: METALIQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022-A02785-38
Record Dates: First submitted 2023-04-25; First posted 2023-05-08 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-08

CONDITIONS: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — Hematologic Tests; Spinal Puncture

STUDY DESIGN:
Intervention Model Description: monocentric, prospective, interventional, exploratory study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- brain metastases from solid cancer (Other): Excision of the cerebral metastasis
  Interventions: Procedure: biological samples (blood test and lumbar puncture)

INTERVENTIONS:
Procedure: biological samples (blood test and lumbar puncture) — On the day of excision of the cerebral metastasis, additional biological samples (blood test and lumbar puncture) will be taken in the operating room.
  A biological sample of the tumor tissue (brain metastases of a solid cancer with contrast uptake of at least 1 cm accessible to surgical excision) will also be taken and preserved by freezing, in accordance with current practice and after obtaining their written agreement. .
  Biological samples (liquid biopsies and tumour) from patients who have explicitly expressed their consent will be kept after the end of the research as part of a biobank in order to be able to carry out any additional analyses.

SUMMARY:
The purpose of the study is to determine in brain metastases and according to feasibility in liquid biopsies:

* Molecular alterations including in particular mutations, amplifications, Copy number gene variants and fusion transcripts identified by high-throughput sequencing;
* The rate of variation either in gain or in loss of expression of the different messenger Ribonucleic Acids by analysis of the transcriptome;
* Epigenetic alterations by methylation of deoxyribonucleic acid clusters by methylome chips.

DETAILED DESCRIPTION:
This is a single-center, prospective, interventional, exploratory study aimed at comparing the molecular alteration profile of liquid biopsies (blood and lumbar puncture) to that of brain metastases.

The population eligible for the study will consist of any patient with cerebral metastases from a solid cancer, at least one of which is accessible to surgical excision.

The study consists of comparing, between brain metastases and liquid biopsies (blood and lumbar puncture), the profiles of genomic, post-genomic and epigenetic alterations as well as the mutational load. To do this, the study only requires a lumbar puncture and a blood test.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over;
* Patient with cerebral metastases from a solid cancer, at least one of which is accessible to surgical excision (contrast enhancement of at least 1 cm);
* Patient able to understand the information related to the study and to read the information leaflet;
* Patient having signed a written informed consent to participate in the study.

Exclusion Criteria:

* Patient with a medical contraindication to surgery and anesthesia;
* Patient whose anatomical location of the cerebral metastasis contraindicates wide resection;
* Patient with a contraindication to performing a lumbar puncture;
* Pregnant, parturient or breastfeeding women;
* Patient participating in another clinical trial, or in a period of exclusion from another clinical trial;
* Patient under guardianship or curatorship, or under a regime of deprivation of liberty;
* Patient not benefiting from a social security scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-06-27 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
molecular alteration profile of liquid biopsies | 1 day
  Compare the molecular alteration profile of liquid biopsies (blood and CSF) to that of brain metastases.
  Will be determined in brain metastases and according to feasibility in liquid biopsies (blood and CSF):
  * Molecular alterations including in particular mutations, amplifications, Copy number gene variants and fusion transcripts identified by high-throughput sequencing ;
  * The rate of variation either in gain or in loss of expression of the different messenger Ribonucleic Acids by analysis of the transcriptome ;
  * Epigenetic alterations by methylation of deoxyribonucleic acid clusters by methylome chips.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Clairval, Marseille, France

IPD SHARING:
Plan to Share IPD: No